CLINICAL TRIAL: NCT04894058
Title: Ureteroscopic Lithotripsy in the Reverse Trendelenburg Position for Upper Ureteral Stones: a Prospective, Randomized, Comparative Study
Brief Title: Ureteroscopic Lithotripsy in the Reverse Trendelenburg Position for Upper Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT2021
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Ureterolithiasis; Ureter Stone; Ureter Calculi
Keywords: Upper ureteral stone; Ureteroscopic lithotripsy; Reverse Trendelenburg
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 ° reverse Trendelenburg (Active Comparator): Patients who underwent ureteroscopic lithotripsy in the 10 ° reverse Trendelenburg position
  Interventions: Procedure: Ureteroscopic lithotripsy
- 20 ° reverse Trendelenburg (Active Comparator): Patients who underwent ureteroscopic lithotripsy in the 20 ° reverse Trendelenburg position
  Interventions: Procedure: Ureteroscopic lithotripsy
- Standard lithotomy (Sham Comparator): Patients who underwent ureteroscopic lithotripsy in standard lithotomy position
  Interventions: Procedure: Ureteroscopic lithotripsy

INTERVENTIONS:
Procedure: Ureteroscopic lithotripsy — After combined spinal and epidural anesthesia, patients were subjected to low pressure perfusion; The semirigid ureteroscope was passed through the urethra to the bladder, after which both ureteral orifices were observed. A 0.035 "soft-tipped guidewire was sent through the ureter orifice and reached the renal pelvis. Subsequently, the patients were placed in the reverse trendelenburg position by leaning 10 ° or 20 ° with their head up and hips down or standard lithotomy position. The ureter stone was accessed with a semirigid ureteroscope. A 273 micron Holmium: yttrium-aluminum-garnet (Ho: YAG) laser was applied as an energy source set at 1.0 J and a speed of 8-10 Hz.

SUMMARY:
This study investigated a previously unassessed operating position for ureteroscopic holmium laser lithotripsy in patients with upper ureteral stone. The reverse Trendelenburg position can reduce migration and improve the stone free rate (SFR). Moreover, less utilization of flexible ureteroscope and hospital stay in reverse Trendelenburg position can reduce the medical cost. Therefore, it can be safely used as an optional surgical method for the treatment of upper ureteral stones.

DETAILED DESCRIPTION:
With the rapid development of urological endoscopy technology, minimally invasive surgery has replaced open surgery in ureteral stones. The majority of upper ureteral stones are treated with endoscopic techniques. In the last 10 years, URSL (Ureteroscopic Lithotripsy) has surpassed SWL (Shock-wave lithotripsy) with its wide use [1]. While URSL was considered in the foreground according to SWL for proximal ureteral stones larger than 1 cm, today it is recommended with equal efficiency and safety with SWL for stones smaller than 1 cm [2]. However, migration of stones to renal calyces is a common problem during ureteroscopic treatment of upper ureteral stones. Migration can be caused by many factors such as the momentum of the laser pulse, stone manipulation of the laser fiber, fluid irrigation pressure and the increase of ureteral dilatation. The degree of migration varies according to the impaction level of the stone and the location in the ureter [3].

The migration of the stone to the renal pelvis and calyces increases the operation time and cost [4-6]. Recently published American Urological Association Guidelines reported that ureteroscopy of ureteral stones performed an average of 1.33 procedures per patient [7]. In order to prevent stone migration, tools have been developed that are used in the proximal of the stone or that interfere with the stone in the kidney after retreatment. Although these developed devices are effective, it has been determined that their additional use causes an additional cost of $ 278 per case as well as extending the operation time [8]. In addition, placing an anti-migration device in the ureter can restrict laser fiber manipulation. Ureterorenoscopes (Flexible URS) that can flex 270 degrees, which can be used to intervene in the stone after retraction into the kidney, have made a very serious improvement, but these devices are not yet available in all centers, especially in developing countries.

There is an in-vitro study using polymer tubes that predict that the proximal ureter should stay higher than the distal ureter in order to prevent retrograde in proximal ureteral stones [9].

ELIGIBILITY:
Inclusion Criteria:

* Obstructive upper ureteral stones

Exclusion Criteria:

* Presence of stent in the ureter at the beginning of the operation
* Serum creatinine value> 1.5 mg / dL
* Pathological ureteral strictures
* Previous open surgery history for the ureteral stone
* Previous pelvic radiotherapy history
* Pregnancy
* Solitary kidney

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of stone migration | One year
  Rate of patients who had a stone migration to renal pelvis or calyces during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santiago JE, Hollander AB, Soni SD, Link RE, Mayer WA. To Dust or Not To Dust: a Systematic Review of Ureteroscopic Laser Lithotripsy Techniques. Curr Urol Rep. 2017 Apr;18(4):32. doi: 10.1007/s11934-017-0677-8. PMID 28271355
- [Background] Drake T, Grivas N, Dabestani S, Knoll T, Lam T, Maclennan S, Petrik A, Skolarikos A, Straub M, Tuerk C, Yuan CY, Sarica K. What are the Benefits and Harms of Ureteroscopy Compared with Shock-wave Lithotripsy in the Treatment of Upper Ureteral Stones? A Systematic Review. Eur Urol. 2017 Nov;72(5):772-786. doi: 10.1016/j.eururo.2017.04.016. Epub 2017 Apr 26. PMID 28456350
- [Background] Elashry OM, Tawfik AM. Preventing stone retropulsion during intracorporeal lithotripsy. Nat Rev Urol. 2012 Dec;9(12):691-8. doi: 10.1038/nrurol.2012.204. Epub 2012 Nov 20. PMID 23165399
- [Background] Cicerello E, Merlo F, Maccatrozzo L. Management of Clinically Insignificant Residual Fragments following Shock Wave Lithotripsy. Adv Urol. 2012;2012:320104. doi: 10.1155/2012/320104. Epub 2012 May 31. PMID 22701479
- [Background] Sea J, Jonat LM, Chew BH, Qiu J, Wang B, Hoopman J, Milner T, Teichman JM. Optimal power settings for Holmium:YAG lithotripsy. J Urol. 2012 Mar;187(3):914-9. doi: 10.1016/j.juro.2011.10.147. Epub 2012 Jan 20. PMID 22264464
- [Background] Pan J, Chen Q, Xue W, Chen Y, Xia L, Chen H, Huang Y. RIRS versus mPCNL for single renal stone of 2-3 cm: clinical outcome and cost-effective analysis in Chinese medical setting. Urolithiasis. 2013 Feb;41(1):73-8. doi: 10.1007/s00240-012-0533-8. Epub 2012 Dec 23. PMID 23532427
- [Background] Segura JW, Preminger GM, Assimos DG, Dretler SP, Kahn RI, Lingeman JE, Macaluso JN Jr. Ureteral Stones Clinical Guidelines Panel summary report on the management of ureteral calculi. The American Urological Association. J Urol. 1997 Nov;158(5):1915-21. doi: 10.1016/s0022-5347(01)64173-9. PMID 9334635
- [Background] Ursiny M, Eisner BH. Cost-effectiveness of anti-retropulsion devices for ureteroscopic lithotripsy. J Urol. 2013 May;189(5):1762-6. doi: 10.1016/j.juro.2012.11.085. Epub 2012 Nov 15. PMID 23159589
- [Background] Patel RM, Walia AS, Grohs E, Okhunov Z, Landman J, Clayman RV. Effect of positioning on ureteric stone retropulsion: 'gravity works'. BJU Int. 2019 Jan;123(1):113-117. doi: 10.1111/bju.14510. Epub 2018 Sep 9. PMID 30098120
- [Derived] Yildiz AK, Doluoglu OG, Kacan T, Keseroglu BB, Ozgur BC, Karakan T. A new position utilizing the effect of gravity in proximal ureteral stones, ureteroscopic lithotripsy in the reverse Trendelenburg position: a prospective, randomized, comparative study. World J Urol. 2023 Dec;41(12):3695-3703. doi: 10.1007/s00345-023-04654-y. Epub 2023 Oct 19. PMID 37855898